CLINICAL TRIAL: NCT05238987
Title: Acute Effect of a Single Dose of Oral Iron on Pancreatic Beta Cell Function in Healthy Individuals: a Quasi-experimental Single Arm Before-and-after (Pre-post) Study
Brief Title: Effect of Taking a Single Tablet of Iron on Insulin Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Padmanaban Venkatesan, Assistant Professor, Department of Biochemistry, Christian Medical College, Vellore, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB min.13294 Dt.26.08.2020
Record Dates: First submitted 2022-02-05; First posted 2022-02-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Insulin Secretion
Keywords: Oral iron; Insulin-Secreting Cells; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Quasi-experimental single arm before-and-after (pre-post) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy men (before-and-after (pre-post) study) (Experimental): Partcipants will undergo a 75g oral glucose tolerance test (OGTT) to document baseline insulin secretion kinetics. One week later, OGTT will be repeated after administering a single dose of ferrous sulphate (120 mg of elemental iron) 2 hours prior to the test.
  Interventions: Dietary Supplement: Ferrous sulphate

INTERVENTIONS:
Dietary Supplement: Ferrous sulphate — Single dose of ferrous sulphate (120 mg of elemental iron)

SUMMARY:
Oral supplementation with highly bioavailable forms of iron, such as ferrous sulphate, is the treatment of choice for iron-deficiency anemia. Iron from ferrous sulphate is efficiently absorbed in the duodenum, resulting in a rapid increase in transferrin saturation and appearance of "free iron" or non-transferrin bound iron (NTBI) in blood. NTBI is highly reactive and can catalyze the generation of reactive oxygen species and cause oxidative tissue damage.

Human pancreatic beta cells are known to express ZIP14, a transporter that has been implicated in uptake of NTBI from blood. In vitro and animal studies have shown that iron loading in beta cells can result in impaired insulin secretion. However, there are no human studies that have looked at the acute effects of oral iron intake on insulin secretion.

In this study, we plan to look at the effect of a single oral dose of ferrous sulphate on insulin secretion kinetics in healthy individuals. A single arm before-and-after (pre-post) study design will be used. Consenting individuals who meet the participation criteria will undergo a 75g oral glucose tolerance test (OGTT) to document baseline insulin secretion kinetics. One week later, OGTT will be repeated after administering a single dose of ferrous sulphate (120 mg of elemental iron) 2 hours prior to the test. Iron-induced change in insulin secretion kinetics will be documented. In addition, we will determine changes in glucose tolerance, insulin resistance and insulin clearance rates.

DETAILED DESCRIPTION:
Oral iron supplementation is the treatment of choice in patients with iron deficiency anemia. In several developing countries, including India, iron is routinely supplemented to pregnant women, especially during the second and third trimesters of pregnancy owing to the increased iron requirement for the placenta and growing fetus.

Oral administration of iron is preferred to intravenous administration because it is effective, relatively cheap and safe. There are many different oral iron preparations and most of them contain iron in the ferrous form (ferrous sulphate, ferrous fumarate, ferrous gluconate, ferrous ascorbate etc.). Although it has been shown that all these preparations are equally effective in increasing hemoglobin levels, ferrous sulphate, being easily available and economical, is the most prescribed iron preparation.

Iron is absorbed in the duodenum. Dietary iron is usually in the ferric form and must be reduced to the ferrous form prior to absorption. This reduction reaction is catalyzed by duodenal ferrireductases (such as duodenal cytochrome b) and is aided by gastric HCl and other reducing substances in the diet, such as vitamin C (ascorbic acid). Administration of iron in the ferrous form (e.g., ferrous sulphate) circumvents this step, thus making it readily bioavailable. Ferrous iron is transported across the luminal membrane of the enterocytes via divalent metal transporter-1 (DMT-1). Iron is then transported across the basolateral membrane (into blood) by another transporter, ferroportin. Hepcidin, a peptide hormone synthesized and secreted by the liver, binds to and degrades ferroportin, thus reducing intestinal iron absorption.

In the blood, iron is transported bound to the plasma protein, transferrin, which binds iron with high affinity. Transferrin is normally saturated to about 30 to 35% of its total iron binding capacity, leaving a large reserve to bind additional iron. In conditions of iron overload, such as hemochromatosis or in patients with thalassemia, transferrin saturation can increase significantly. When transferrin saturation increases beyond 60% and especially as it approaches 80%, a small but significant amount of iron circulates in blood that is not bound to transferrin. This fraction, called "labile iron" or non-transferrin bound iron (NTBI), is highly reactive and can cause oxidative tissue damage.

NTBI is rapidly cleared from circulation, mainly by hepatocytes. It has been shown that ZIP14 is physiologically the most important transporter that transports NTBI into hepatocytes. Recently, it was shown that ZIP14 is also expressed on human pancreatic beta cells and that it may mediate NTBI uptake by these cells. Several in vitro and animal studies have shown that iron overload impairs pancreatic beta cell function. Patients with hemochromatosis are known to accumulate iron in the beta cells, resulting in diabetes due to decreased insulin secretory capacity. On the other hand, iron chelation or dietary iron restriction improves insulin secretion in mouse models of diabetes. Similarly, iron chelation in hemochromatosis and thalassemia also improved insulin secretion. These studies prove a strong link between increased iron and impaired beta cell function.

It has been shown that, following a single dose of ferrous sulphate (containing 60-100 mg of elemental iron), transferrin saturation increases rapidly and peaks (at ~ 80%) 2 hours after administration. This is associated with a significant increase in NTBI, which also peaks at 2 hours. Given that oral iron administration increases NTBI in blood and that pancreatic beta cells take up NTBI via ZIP14, we hypothesized that oral iron may lead to increased beta cell iron levels which may then cause impaired insulin secretion

In order to test this hypothesis, we plan to conduct a quasi-experimental single arm before-and-after study, where insulin secretion kinetics will be determined at baseline and after a single dose of iron (ferrous sulphate, 120 mg elemental iron) in healthy men.

Healthy male volunteers will be recruited from among the staff of Christian Medical College, Vellore after obtaining written informed consent.Participants will undergo a 75g oral glucose tolerance tests (OGTT) to document baseline insulin secretion kinetics. One week later, the OGTT will be repeated after a single dose of ferrous sulphate (120 mg of elemental iron) given 2 hours before the test. Serum levels of glucose, insulin, C-peptide, serum iron and transferrin saturation will be measured during both OGTT. The effects of iron on insulin secretion kinetics will be documented. In addition, we will determine if changes occur in glucose tolerance, insulin resistance and insulin clearance rates.

ELIGIBILITY:
Inclusion Criteria:

BMI - 18 to 30 kg/m^2

Exclusion Criteria:

1. Known case of diabetes mellitus/pre-diabetes
2. History of chronic inflammatory disease
3. Anemia (detection of pallor on examination). Absence of anemia will be confirmed by hemoglobin estimation done at the time of baseline OGTT based on WHO criteria.
4. On iron supplementation
5. History of any gastrointestinal disorders that might affect absorption of iron/glucose

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Change in insulin secretion kinetics | 2 hours from intake of 120 mg of elemental iron
  Change in insulin secretion rate as determined by deconvolution of C-peptide levels in blood during an oral glucose tolerance test based on a previously published mathematical model (Van Cauter et al., 1992).
Change in disposition index | 2 hours from intake of 120 mg of elemental iron
  Disposition index is a measure of beta-cell function which is calculated as a product of insulin sensitivity and insulin secretion during an oral glucose tolerance test
Change in insulinogenic index | 2 hours from intake of 120 mg of elemental iron
  A measure of beta-cell function which calculates the increase in insulin secretion in response to increase in glucose concentration during an oral glucose tolerance test

SECONDARY OUTCOMES:
Change in glucose tolerance | 2 hours from intake of 120 mg of elemental iron
  Glucose tolerance will be determined by calculating the area under the curve (AUC) of glucose levels during oral glucose tolerance test
Change in insulin sensitivity | 2 hours from intake of 120 mg of elemental iron
  Insulin sensitivity which is a measure of insulin action will be calculated using the Matsuda index (Matsuda and DeFronzo, 1999)
Change in insulin clearance rate | 2 hours from intake of 120 mg of elemental iron
  Insulin clearance rate which is a measure of rate of disappearance of insulin from the blood will be calculated as described previously (Castillo et al., 1994)

CONTACTS AND LOCATIONS:
Overall Officials: Padmanaban Venkatesan, M.D., Principal Investigator — Christian Medical College, Vellore, India; Joe Varghese, M.D.,PhD, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham D, Rogers J, Gault P, Kushner JP, McClain DA. Increased insulin secretory capacity but decreased insulin sensitivity after correction of iron overload by phlebotomy in hereditary haemochromatosis. Diabetologia. 2006 Nov;49(11):2546-51. doi: 10.1007/s00125-006-0445-7. Epub 2006 Sep 22. PMID 17019598
- [Background] Auerbach M, Adamson JW. How we diagnose and treat iron deficiency anemia. Am J Hematol. 2016 Jan;91(1):31-8. doi: 10.1002/ajh.24201. Epub 2015 Nov 17. PMID 26408108
- [Background] Backe MB, Moen IW, Ellervik C, Hansen JB, Mandrup-Poulsen T. Iron Regulation of Pancreatic Beta-Cell Functions and Oxidative Stress. Annu Rev Nutr. 2016 Jul 17;36:241-73. doi: 10.1146/annurev-nutr-071715-050939. Epub 2016 May 4. PMID 27146016
- [Background] Brissot P, Ropert M, Le Lan C, Loreal O. Non-transferrin bound iron: a key role in iron overload and iron toxicity. Biochim Biophys Acta. 2012 Mar;1820(3):403-10. doi: 10.1016/j.bbagen.2011.07.014. Epub 2011 Aug 9. PMID 21855608
- [Background] Castillo MJ, Scheen AJ, Letiexhe MR, Lefebvre PJ. How to measure insulin clearance. Diabetes Metab Rev. 1994 Jul;10(2):119-50. doi: 10.1002/dmr.5610100205. No abstract available. PMID 7956676
- [Background] Coffey R, Knutson MD. The plasma membrane metal-ion transporter ZIP14 contributes to nontransferrin-bound iron uptake by human beta-cells. Am J Physiol Cell Physiol. 2017 Feb 1;312(2):C169-C175. doi: 10.1152/ajpcell.00116.2016. Epub 2016 Nov 30. PMID 27903581
- [Background] Cooksey RC, Jones D, Gabrielsen S, Huang J, Simcox JA, Luo B, Soesanto Y, Rienhoff H, Abel ED, McClain DA. Dietary iron restriction or iron chelation protects from diabetes and loss of beta-cell function in the obese (ob/ob lep-/-) mouse. Am J Physiol Endocrinol Metab. 2010 Jun;298(6):E1236-43. doi: 10.1152/ajpendo.00022.2010. Epub 2010 Mar 30. PMID 20354157
- [Background] Dresow B, Petersen D, Fischer R, Nielsen P. Non-transferrin-bound iron in plasma following administration of oral iron drugs. Biometals. 2008 Jun;21(3):273-6. doi: 10.1007/s10534-007-9116-5. Epub 2007 Sep 13. PMID 17851733
- [Background] Farmaki K, Angelopoulos N, Anagnostopoulos G, Gotsis E, Rombopoulos G, Tolis G. Effect of enhanced iron chelation therapy on glucose metabolism in patients with beta-thalassaemia major. Br J Haematol. 2006 Aug;134(4):438-44. doi: 10.1111/j.1365-2141.2006.06203.x. Epub 2006 Jul 4. PMID 16822284
- [Background] Fuqua BK, Vulpe CD, Anderson GJ. Intestinal iron absorption. J Trace Elem Med Biol. 2012 Jun;26(2-3):115-9. doi: 10.1016/j.jtemb.2012.03.015. Epub 2012 May 8. PMID 22575541
- [Background] Geisser P, Burckhardt S. The pharmacokinetics and pharmacodynamics of iron preparations. Pharmaceutics. 2011 Jan 4;3(1):12-33. doi: 10.3390/pharmaceutics3010012. PMID 24310424
- [Background] Goddard AF, James MW, McIntyre AS, Scott BB; British Society of Gastroenterology. Guidelines for the management of iron deficiency anaemia. Gut. 2011 Oct;60(10):1309-16. doi: 10.1136/gut.2010.228874. Epub 2011 May 11. PMID 21561874
- [Background] Hansen JB, Tonnesen MF, Madsen AN, Hagedorn PH, Friberg J, Grunnet LG, Heller RS, Nielsen AO, Storling J, Baeyens L, Anker-Kitai L, Qvortrup K, Bouwens L, Efrat S, Aalund M, Andrews NC, Billestrup N, Karlsen AE, Holst B, Pociot F, Mandrup-Poulsen T. Divalent metal transporter 1 regulates iron-mediated ROS and pancreatic beta cell fate in response to cytokines. Cell Metab. 2012 Oct 3;16(4):449-61. doi: 10.1016/j.cmet.2012.09.001. Epub 2012 Sep 20. PMID 23000401
- [Background] Jenkitkasemwong S, Wang CY, Coffey R, Zhang W, Chan A, Biel T, Kim JS, Hojyo S, Fukada T, Knutson MD. SLC39A14 Is Required for the Development of Hepatocellular Iron Overload in Murine Models of Hereditary Hemochromatosis. Cell Metab. 2015 Jul 7;22(1):138-50. doi: 10.1016/j.cmet.2015.05.002. Epub 2015 May 28. PMID 26028554
- [Background] Kapil U, Kapil R, Gupta A. National Iron Plus Initiative: Current status & future strategy. Indian J Med Res. 2019 Sep;150(3):239-247. doi: 10.4103/ijmr.IJMR_1782_18. PMID 31719294
- [Background] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Background] McClain DA, Abraham D, Rogers J, Brady R, Gault P, Ajioka R, Kushner JP. High prevalence of abnormal glucose homeostasis secondary to decreased insulin secretion in individuals with hereditary haemochromatosis. Diabetologia. 2006 Jul;49(7):1661-9. doi: 10.1007/s00125-006-0200-0. Epub 2006 Mar 15. PMID 16538487
- [Background] Nemeth E, Tuttle MS, Powelson J, Vaughn MB, Donovan A, Ward DM, Ganz T, Kaplan J. Hepcidin regulates cellular iron efflux by binding to ferroportin and inducing its internalization. Science. 2004 Dec 17;306(5704):2090-3. doi: 10.1126/science.1104742. Epub 2004 Oct 28. PMID 15514116
- [Background] Solomon TPJ. Sources of Inter-individual Variability in the Therapeutic Response of Blood Glucose Control to Exercise in Type 2 Diabetes: Going Beyond Exercise Dose. Front Physiol. 2018 Jul 13;9:896. doi: 10.3389/fphys.2018.00896. eCollection 2018. PMID 30061841
- [Background] Van Cauter E, Mestrez F, Sturis J, Polonsky KS. Estimation of insulin secretion rates from C-peptide levels. Comparison of individual and standard kinetic parameters for C-peptide clearance. Diabetes. 1992 Mar;41(3):368-77. doi: 10.2337/diab.41.3.368. PMID 1551497
- [Background] Blesia V, Patel VB, Al-Obaidi H, Renshaw D, Zariwala MG. Excessive Iron Induces Oxidative Stress Promoting Cellular Perturbations and Insulin Secretory Dysfunction in MIN6 Beta Cells. Cells. 2021 May 9;10(5):1141. doi: 10.3390/cells10051141. PMID 34065122
- [Derived] Venkatesan P, Ramasamy J, Vanitha S, Jacob M, Varghese J. Impaired pancreatic beta-cell function after a single dose of oral iron: A before-and-after (pre-post) study. J Hum Nutr Diet. 2023 Jun;36(3):1111-1120. doi: 10.1111/jhn.13074. Epub 2022 Sep 7. PMID 36000222